CLINICAL TRIAL: NCT03091114
Title: Predictive Factors for Failure of Internal Fixations of Lower Limb Fractures: a Prospective Cohort Study
Brief Title: Predictive Factors for Failure of Internal Fixations of Lower Limb Fractures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Tim Mathes, Principal Investigator, University of Witten/Herdecke
Other Study IDs: V01-A0
Record Dates: First submitted 2017-03-13; First posted 2017-03-27 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Lower Limb Fractures
Keywords: fractures, risk prediction
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

A predictive factor is a measure that predicts treatment response. Decisions on internal fixations of lower limb fractures should regard predictive factors to personalize (e.g. age) treatment. However for most potentially influencing factors valid data on the predictive value is sparse.

Objectives:

The objective of this study is to identify predictive factors and quantify their predictive ability for treatment failure in patients with limb fractures treated with osteosynthesis.

Methods:

Patients Adult patients (≥18 year) with isolated fractures scheduled for urgent or semi-urgent surgery using internal fixations because of lower limb fractures.

The predictive value of the following exposures will be analyzed:

* Age
* Gender
* Diabetes
* Smoking status
* Body Mass Index
* Open fractures
* Peripheral arterial disease

Outcome The outcome will be (time to) reoperation of the same fracture because of failure of internal fixation due to nonunion or implant failure.

Study design A prospective observational cohort study will be performed. Sample size 300 patients will be included.

Statistical analysis:

For the main analysis a multivariate stratified Cox proportional hazard model will be used. The Model will be stratified according to the indication. In the Cox proportional hazard model all predictive factors will be entered simultaneously to quantify the independent influence (adjusted for all other factors) of each factor. The strength of prediction will be described with hazard rations and their corresponding 95% confidence intervals.

DETAILED DESCRIPTION:
see study protocol: https://uni-wh.de/fileadmin/user_upload/03_G/07_Humanmedizin/05_Institute/IFOM/IFF-PROFAK_Protocol.pdf

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years) with isolated fractures scheduled for urgent or semi-urgent surgery using internal fixations because of the following lower limb fractures will be included:

* Tibia fractures
* Femur fractures
* Ankle fractures
* Calcaneal fractures

Exclusion Criteria:

* Periprosthetic fractures
* Insufficient knowledge of the German language
* Strong cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower limb fractures.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure of internal fixation | 6 months +/- 2 weeks (survival analysis)
  Failure of internal fixation due to nonunion or implant failure

SECONDARY OUTCOMES:
Pain | 6 months +/- 2 weeks
  Pain numerical rating scale (NRS) >3
Physical functioning | 6 months +/- 2 weeks
  E.g. climbing stairs

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mathes, Dr., Principal Investigator — University of Witten/Herdecke
Locations (1):
- Clinic for orthopedics, trauma surgery and sports traumatology, hospital Cologne Merheim, Cologne, North-Rhine-Westfalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
All data on predictive factors and outcomes will be made available. Published as supplemental material open access (anticipated 12/2018).

REFERENCES:
- [Derived] Prediger B, Tjardes T, Probst C, Heu-Parvaresch A, Glatt A, Dos Anjos DR, Bouillon B, Mathes T. Factors predicting failure of internal fixations of fractures of the lower limbs: a prospective cohort study. BMC Musculoskelet Disord. 2021 Sep 16;22(1):798. doi: 10.1186/s12891-021-04688-6. PMID 34530793